CLINICAL TRIAL: NCT04849247
Title: 68Ga-DOTA-FAPI and 177Lu-DOTA-FAPI Theranostic Pair in Patients With Various Types of Cancer (Locally Advanced or Metastatic Cancer)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XMYYL2021KYSB082
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: 177Lu-DOTA-FAPI; 68Ga-DOTA-FAPI; Theranostic

STUDY DESIGN:
Intervention Model Description: This is a first-in-human 3 + 3 study design to identify dose limiting toxicity and recommended phase 2 dose Masking: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 177Lu-DOTA-FAPI dose escalation therapy study (Experimental): Patients will be undergo 68Ga-DOTA-FAPI PET/CT scans to confirm eligibility for the 177Lu-DOTA-FAPI therapy. Patients with sufficient lesion uptake of 68Ga DOTA-FAPI PET/CT will be offered therapy. Escalating doses of 30-150 mCi of 177Lu-DOTA-FAPI will be administered in a traditional 3+3 dose escalation design. After escalation, 10 additional patients will be enrolled into a dose expansion cohort.
  Interventions: Drug: 68Ga-DOTA-FAPI, 177Lu-DOTA-FAPI
- Recommended Phase 2 dose 177Lu-DOTA-FAPI therapy study (Experimental): Patients will be undergo 68Ga-DOTA-FAPI PET/CT scans to confirm eligibility for the 177Lu-DOTA-FAPI therapy. 10 patients will be enrolled in the dose expansion cohort and received the highest dose achieved in the 177Lu-DOTA-FAPI dose escalation therapy study
  Interventions: Drug: 68Ga-DOTA-FAPI, 177Lu-DOTA-FAPI

INTERVENTIONS:
Drug: 68Ga-DOTA-FAPI, 177Lu-DOTA-FAPI — PET imaging using 68Ga-DOTA-FAPI will be used to diagnose patients who are eligible for treatment with the 177Lu-DOTA-FAPI.

SUMMARY:
This is a Phase I, first-in-human study to evaluate the safety and efficacy of the 68Ga-DOTA-FAPI and 177Lu-DOTA-FAPI theranostic pair in patients with various types of cancer (locally advanced or metastatic cancer).

DETAILED DESCRIPTION:
This is a Phase I, first-in-human study to evaluate the safety and efficacy of the 68Ga-DOTA-FAPI and 177Lu-DOTA-FAPI theranostic pair in patients with various types of cancer. PET imaging using 68Ga-DOTA-FAPI will be used to diagnose patients who are eligible for the 177Lu-DOTA-FAPI. The overall purpose of this study is to identify the dose limiting toxicity (DLT) and recommended phase 2 dose (RP2D) of 177Lu-DOTA-FAPI. A 3+3 study design in is proposed to identify the RP2D of 177Lu-DOTA-FAPI. An expansion group will receive the RP2D in order to obtain initial estimates of response and additional information on safety of 177Lu-DOTA-FAPI.

The hypotheses of this phase I study are that a) 68Ga-DOTA-FAPI will detect lesions in patients with various types of locally advanced or metastatic cancer. b) the theranostic pair 68Ga-DOTA-FAPI and 177Lu-DOTA-FAPI will be safe and well tolerated c) we will be able to identify a Recommended Phase 2 Dose (RP2D) for 177Lu-DOTA-FAPI therapy to be used in subsequent Phase II trials.

ELIGIBILITY:
Inclusion Criteria:

* [68Ga]Ga-DOTA-FAPI PET/CT Inclusion Criteria: (i) adult participants (aged 18 years or order); (ii) Confirmed presence of various types of locally advanced or metastatic cancer with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis); (iii) Participant must have documented tumor progression during or following at least one prior systemic regimen as established by CT or MRI scan within 28 days of enrollment; (iv) participants who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee. (v) Eastern Cooperative Oncology Group Performance Status ≤ 2; (vi) Participant must have completed prior therapy at least 1 month (washout period) prior to [68Ga]Ga DOTA-FAPI PET scan. Any clinically significant toxicity (with the exceptions of hair loss and sensory neuropathy) related to prior therapy resolved to Grade 1 or baseline;
* Hematologic parameters defined as:

  (i)Absolute neutrophil count (ANC) ≥ 1000 cells/mm3; (ii)Platelet count ≥ 100,000/mm3; (iii)Hemoglobin ≥ 8 g/dL;
* Blood chemistry levels defined as:

  (i) AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN); (ii) Total bilirubin ≤ 2 times ULN; (iii) Creatinine ≤ 2 times ULN; (iv) Anticipated life expectancy ≥ 6 months; (v) Able to remain motionless for up to 10-20 minutes per scan;
* [177Lu]Lu-DOTA-FAPI therapy Inclusion Criteria: (i) Completion of entry into [68Ga]Ga-DOTA-FAPI PET study and completion of scan; (ii) CThe presence of at least one measurable disease by [68Ga]Ga-DOTA-FAPI PET/CT (SUVmax > 10-fold above normal lung or liver);
* Exclusion Criteria:

  (i) 1.Participant on any chemical anticoagulant including antiplatelet agents (excluding ASA); (ii)Participants with Class 3 or 4 NYHA Congestive Heart Failure (iii) Clinically significant bleeding within two weeks prior to trial entry (e.g. gastrointestinal bleeding, intracranial bleeding); (iv) Pregnant or lactating women; (v)Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e. larger than what is required for placement of a central venous access, percutaneous feeding tube, or biopsy) within 28 days prior to study day 1 or anticipated surgery within the subsequent 6 weeks; (vi)Has an additional active malignancy requiring therapy within the past 2 years; (vii)Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy; (viii)Psychiatric illness/social situations that would interfere with compliance with study requirements; (ix)Cannot undergo PET/CT scanning because of weight limits (350 lbs); (x)INR>1.2; PTT>5 seconds above UNL

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
68Ga-DOTA-FAPI PET/CT imaging | 1 hours from time of injection
  Assessment of 68Ga-DOTA-FAPI PET/CT imaging to detect lesions in patients with various types of cancer (locally advanced or metastatic cancer)
[177Lu]Lu-DOTA-FAPI dose escalation therapy | 60 days from time of injection
  Frequency of dose-limiting toxicities (DLT) of 177Lu-DOTA-FAPI at escalating dose levels of 177Lu-DOTA-FAPI

SECONDARY OUTCOMES:
Assessment of organ dosimetry of 177Lu-DOTA-FAPI | 1-7 days from time of injection
  Assessment of organ dosimetry of 177Lu-DOTA-FAPI using SPECT/CT imaging at various timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- First affiliated hospital of xiamen university, Xiamen, Fujian, China